CLINICAL TRIAL: NCT03299920
Title: Opioid Consumption After Knee Arthroscopy With and Without the Use of New Standardized Patient/Family Instructions for Postoperative Analgesic Use
Brief Title: Opioid Consumption After Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giorgio Veneziano (Other)
Responsible Party: Sponsor-Investigator, Giorgio Veneziano, Director, Regional Anesthesia Service, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00710
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Surgical Procedure, Unspecified; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients will receive standardized instruction from a study nurse, tailored to understanding pain management after nerve blocks and maximizing utilization of non-opioid analgesics.
  Interventions: Other: Standardized instructions
- Control (Other): Patient will receive conventional instructions on postoperative pain management.
  Interventions: Other: Conventional instructions

INTERVENTIONS:
Other: Standardized instructions — Specific instructions related to peripheral nerve block.
  Arms: Intervention
Other: Conventional instructions — Usual post-operative instructions.
  Arms: Control

SUMMARY:
This is a prospective, randomized trial of patients undergoing outpatient knee arthroscopy surgery and receiving a peripheral nerve block. Patients will be randomized to either receive standard discharge teaching or specialized teaching regarding pain control following a nerve block. Patients will be asked to complete a journal for 5 days recording their pain scores, opioid medication usage, and overall satisfaction with pain control at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient of age less than 20 years presenting to NCH main campus for knee arthroscopy
* American Society of Anesthesiology physical status I or II

Exclusion Criteria:

* Anterior cruciate ligament repair or reconstruction
* Admission to hospital
* Inability or refusal to receive femoral nerve blockade
* Body mass index > 99 percentile
* Hydrocodone allergy or intolerance
* Acetaminophen allergy or intolerance
* Non-steroidal anti-inflammatory allergy or intolerance
* Pregnancy
* Interpreter requirement
* Opioid use within 3 months prior to surgery
* Previous knee surgery at WSC after Jan. 1, 2017
* History of opioid abuse or dependence

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Number of opioid medication doses taken | Post-op day 5

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Veneziano, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No